CLINICAL TRIAL: NCT00899340
Title: Protein Expression Profiles in Oropharyngeal Squamous Cell Carcinoma
Brief Title: Protein Expression in Tumor Tissue Samples From Patients With Cancer of the Oropharynx
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Murphy, MD, Professor of Medicine, Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC HN 0624; VU-VICC-HN-0624; VU-VICC-IRB-060380
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Gene Expression Profiling; Microarray Analysis; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: gene expression analysis — profiles of HPV(+) and (-) HNSCCs
Genetic: microarray analysis — microarray analysis
  Other Names: SAM - significance Analysis of microarrays
Genetic: protein expression analysis — protein expression analysis
Other: immunohistochemistry staining method — immunohistochemistry staining method
Other: laboratory biomarker analysis — laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying the proteins expressed in samples of tumor tissue from patients with cancer may help doctors identify and learn more about biomarkers related to cancer. It may also help doctors plan better treatment for patients with cancer of the oropharynx.

PURPOSE: This laboratory study is looking at protein expression in tumor tissue samples from patients with cancer of the oropharynx.

DETAILED DESCRIPTION:
OBJECTIVES:

* To investigate if some of the differences in gene expression are also reflected at the protein level.
* To determine whether differences in gene expression that are also reflected at the protein level can be used to develop markers for early detection and disease surveillance.
* To identify targets for therapy.

OUTLINE: Archived tumor tissue samples are analyzed for expression of standard immunohistological markers (e.g., p16, p53, and Ki-67) as well as expression of genes identified in a previous gene expression study. Protein expression data are tested for clinical and demographic correlates and compared with gene expression data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of squamous cell carcinoma of the oropharynx
* Tumor tissue samples available from Vanderbilt Head and Neck Tumor Repository and Vanderbilt Pathology archives

Exclusion Criteria:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2006-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Development of biomarkers for early detection or recurrence surveillance | after 7 months of tissue collection
Identification of therapeutic targets and individualization of treatment based on the biology of squamous cell carcinoma of the oropharynx | after 7months of tissue collection

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Murphy, MD, Study Chair — Vanderbilt-Ingram Cancer Center